CLINICAL TRIAL: NCT06271915
Title: Effect of Cervical Spine Mobilization With Movement on Lateral Epicondylitis: A Randomized Controlled Trial.
Brief Title: Role of Cervical Spine Mobilization on Lateral Epicondylitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed ElMelhat, Assisatnt Professor of Phyiscal Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: cervical spine mobilization
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Lateral Epicondylitis
Keywords: Tennis Elbow, Elbos tendinitis, Cervical Spine, Manual Therapy.; Central sensitization
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lateral epicondilitis with SNAG's (Experimental): The intervention group, will receive mulligan's technique on C4-C7 cervical region and eccentric exercises to the affected forearm interventions done 2 times per week, 45 minutes each session for 4 weeks
  Interventions: Other: SNAGs - eccentric exercise
- lateral epicondylitis (Active Comparator): control group will receives only localized treatment as eccentric exercise, stretching of forearm extensors, cross-friction massage and ultrasound with frequency 3 MHz and intensity 2 W/cm2, 100% duty cycle on the affected forearm.
  interventions done 2 times per week, 45 minutes each session for 4 weeks
  Interventions: Other: SNAGs - eccentric exercise

INTERVENTIONS:
Other: SNAGs - eccentric exercise — intervention done 2 times per week, 45 minutes each session for 4 weeks

SUMMARY:
The study's primary goal is to examine the effectiveness of Mulligan's technique in reducing hyperalgesia in lateral epicondylitis, focusing on cervical spine, while also investigating its influence on central sensitization in relation to lateral epicondylitis.

DETAILED DESCRIPTION:
Lateral epicondylitis (LE) also known as tennis elbow, results from an overuse injury due to eccentric overload on the common extensor tendon, particularly at the origin of the extensor carpi radialis brevis (ECRB). This condition is frequently triggered by repetitive strain during tasks involving repeated gripping and loaded wrist extension. Lateral epicondylitis affects 1% to 3% of population, especially in middle-aged people. In addition, patients with LE suffer from pain or burning on the common extensor origin of the forearm that may radiate into the upper arm or downward to the forearm. The pain can be exacerbated with resisted wrist extension, forearm supination and middle finger extension. The initial approach to manage lateral epicondylitis involves conservative therapy, including eccentric training, stretching and local manual therapy.

In individuals with lateral epicondylitis, the experience of mechanical hyperalgesia characterized by increased pain sensitivity during cold application is indicative of potential central sensitization. Central sensitization involves heightened reactivity of nociceptors within the central nervous system, resulting in increased responsiveness to both normal and sub-threshold afferent input. This heightened sensitivity also includes increased responsiveness to non-noxious stimuli and an elevated pain response triggered by stimuli originating outside the area of injury, indicating an expanded receptive field. Furthermore, cervical dysfunction is observable in individuals with LE even in the absence of neck pain indicating the involvement of central sanitization. The potential influence of cervical manual therapy on reducing mechanical hyperalgesia aligns with addressing central sensitization, contributing to a comprehensive approach in managing pain and sensitivity associated with lateral epicondylitis.

Its hypothesized that spinal manual therapy on the cervical spine is likely to yield positive short-term outcomes on pain-free grip and the pain threshold elicited by pressure over the lateral humeral epicondyle. As the mechanism of manual techniques proves effective on mechanical, neurophysiological, and peripheral receptors while inducing supraspinal pain inhibition related with sympathoexcitation3, hypoalgesia could occur following the application of these techniques.

Mulligan's mobilization and SNAGS approach involves applying force and direction to the facet joint, reaching the end range of motion. This technique aims to restore the original position of cervical spine facet joint which possibly impacts the hyperalgesia frequently associated with lateral epicondylitis. Moreover, mobilization with movement induces biomechanical changes in the vertebrae, affecting central processing. It restrains pain mechanisms, reduces neck dysfunction, and improves neck disability.

Notably, previous studies investigated, that they have indicated the need for further research to determine the effects of spinal manipulation on hypoalgesia. Furthermore, other study previously explored the effects of manual therapy on the thoracic spine concerning pain-free grip and sympathetic activity in patients with lateral epicondylitis producing favorable outcomes needing additional exploration when including the cervical spine.

As such, the main objective of this study is to evaluate Mulligan's technique effectiveness in relieving mechanical and cold hyperalgesia in individuals with lateral epicondylitis, with a specific emphasis on the cervical spine region. Additionally, the research aims to investigate the impact of Mulligan's technique on central sensitization in the cervical spine and its influence on lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* a positive Maudsley's test and Cozen's test,
* positive Spurling and axial distraction tests
* limited range of motion of the cervical spine
* a positive upper limb tension test (ULTT)
* middle-aged individuals (40-60 years old).

Exclusion Criteria:

* participants with any pathologies
* participants involved in other studies
* patients undergoing corticosteroids treatment
* physical therapy sessions, or surgical interventions for elbow or cervical spine issues within the past year
* individuals afflicted by inflammatory, infectious, or systematic diseases
* participants experiencing bilateral elbow pain or tumor diseases are excluded.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Leeds assessment of neuropathic symptoms and sign (LANSS) scale | Baseline
  is a questionnaire to screen neuropathic pain. It Contains five items concerning self-reported pain symptoms, and two items depending on simple clinical examination provided by healthcare professional that's targeting pin-prick threshold and allodynia. Scoring with LANSS: if the participant gains 12 or more out of 24, the pain will be considered of neuropathic origin. LANSS scale demonstrated a sensitivity (83%) and specificity of (87%), effectively identifying (85%) of neuropathic pain.
Pain-free hand grip test | Baseline
  Pain-free grip test is a reliable and valid tool to use with lateral epicondylitis patients with using dynamometer to measure the grip force applied to the point of pain. Some studies recommended to perform the test with elbow relaxed extended, forearm pronated, and repeated 3 times with 1 minute interval, then comparing the average of 3 measurements between affected and non-affected.

SECONDARY OUTCOMES:
The Numeric Rating Scale (NRS) | baseline
  The Numeric Rating Scale (NRS) is a reliable and valid instrument for assessing pain intensity in chronic cases, as evidenced by its effective adaptation into an Arabic version: Arabic Numeric Pain Rating Scale (ANPRS). Reliability of the ANPRS (ICC 0.89) considered good to excellent. Arabic version of NRS considered reliable and valid tool to measure pain levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient physical therapy, Faculty of physical therapy, Giza, Egypt

REFERENCES:
- [Result] Coombes BK, Bisset L, Vicenzino B. Management of Lateral Elbow Tendinopathy: One Size Does Not Fit All. J Orthop Sports Phys Ther. 2015 Nov;45(11):938-49. doi: 10.2519/jospt.2015.5841. Epub 2015 Sep 17. PMID 26381484
- [Result] Cleland JA, Whitman JM, Fritz JM. Effectiveness of manual physical therapy to the cervical spine in the management of lateral epicondylalgia: a retrospective analysis. J Orthop Sports Phys Ther. 2004 Nov;34(11):713-22; discussion 722-4. doi: 10.2519/jospt.2004.34.11.713. PMID 15609491